CLINICAL TRIAL: NCT02575339
Title: An Open Label Randomized Phase I/II Trial of MLN0128 Compared to Sorafenib in Patients With Advanced or Metastatic Hepatocellular Carcinoma: Big Ten Cancer Research Consortium BTCRC-GI13-002
Brief Title: MLN0128 Compared to Sorafenib in Advanced or Metastatic Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funder Decision
Sponsor: Kathy Miller (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); Big Ten Cancer Research Consortium (Other)
Responsible Party: Sponsor-Investigator, Kathy Miller, Sponsor-Investigator, Big Ten Cancer Research Consortium
Organization: Big Ten Cancer Research Consortium (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTCRC GI13-002
Record Dates: First submitted 2015-10-09; First posted 2015-10-14 (Estimated); Results first posted 2022-03-31 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer; HCC
Keywords: MLN0128; Sapanisertib; TORC1/2 inhibitor; INK128; Nexavar; Sorafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — sapanisertib; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase I MLN0128 Dose Escalation Study (Experimental): Subjects will receive MLN0128 orally on days 1, 8, 15 and 22 in successive cohorts.
  Cohort 1 MLN0128 15mg each week (QW); Cohort 2 MLN0128 20mg QW; Cohort 3 MLN0128 30mg QW
  Interventions: Drug: MLN0128
- Phase II Arm A: MLN0128 (Experimental): Subjects randomized to experimental arm will receive MLN0128 orally at the recommended phase II dose (RP2D) once weekly.
  Interventions: Drug: MLN0128 (RP2D)
- Phase II Arm B: Sorafenib (Active Comparator): Subjects randomized to control arm will receive sorafenib 400mg by mouth (PO) twice a day (BID) daily.
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: MLN0128 — Phase I Dose Escalation Study Cohort 1 MLN0128 15mg QW; Cohort 2 MLN0128 20mg QW; Cohort 3 MLN0128 30mg QW
  Other Names: Sapanisertib
  Arms: Phase I MLN0128 Dose Escalation Study
Drug: MLN0128 (RP2D) — Phase II Arm A:
  MLN0128 administered orally at the recommended phase II dose (RP2D) once weekly.
  Other Names: Sapanisertib
  Arms: Phase II Arm A: MLN0128
Drug: Sorafenib — Phase II Arm B:
  Sorafenib administered at 400mg PO BID daily
  Other Names: Nexavar
  Arms: Phase II Arm B: Sorafenib

SUMMARY:
This is an open label, multi-center, randomized phase I/II study of MLN0128 versus standard sorafenib. Eligible subjects in the phase I trial will receive MLN0128 in escalating doses. Eligible subjects in the phase II trial will be 1:1 randomized to either the MLN0128 arm or the sorafenib arm.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center trial.

The phase 1 dose escalation trial will evaluate MLN0128 in a standard 3+3 successive cohort design to identify the highest planned dose level. Phase II trial subjects will be 1:1 randomized to receive either MLN0128 (investigational arm) or sorafenib (control arm).

PHASE I DOSE ESCALATION INVESTIGATIONAL TREATMENT:

Cohort 1 (dose level +1) will consist of 3-6 evaluable patients who will receive MLN0128 15mg on day 1 of the 28-day cycle.

Cohort 2 (dose level +2) will consist of 3-6 evaluable patients who will receive MLN0128 20mg on day 1 of the 28-day cycle.

Cohort 3 (dose level +3) will consist of 3-6 evaluable patients who will receive MLN0128 30mg on day 1 of the 28-day cycle.

Subjects will be evaluated for dose limiting toxicity (DLT) in the first 28 days of treatment (1 cycle). However, decisions to move to next dose escalation cohort will not be made until all subjects complete 2 cycles of therapy at a given dose. There will be no further dose escalation beyond dose level +3.

PHASE II INVESTIGATIONAL TREATMENT:

Randomization will take place following completion of the screening evaluations and eligibility assessments. Stratification factors will be employed during randomization to minimize between-arm assignment imbalance.

* 1 Child-Pugh score 5-6
* 2 Child-Pugh score 7

Within the strata, subjects will be randomly assigned with equal probability to either the investigational arm (Arm A: MLN0128) or the control arm (Arm B: sorafenib).

Arm A: MLN0128 will be administered orally at the recommended phase II dose (RP2D) once weekly.

Arm B: Sorafenib will be administered at 400mg PO BID daily, with dose adjustment per standard of care.

A new treatment cycle (1 cycle = 28 days) will only be initiated when all of the following conditions are met:

* Absolute neutrophil count (ANC) ≥ 1.5 x 10*9/L
* Platelets ≥ 50 x 10*9/L
* Non-hematologic treatment related toxicities have improved to grade 1 or resolved per Common Terminology Criteria for Adverse Events v4.0 (CTCAE)

Treatment may continue until progression, unacceptable toxicity, or withdrawal from study.

Estimated Life Expectancy: ≥ 3 months

Subjects must have adequate organ function, as specified below, within 7 days before study registration:

Bone marrow reserve consistent with:

* Absolute neutrophil count (ANC) ≥ 1.5 x 10*9/L
* Platelet count ≥ 50 x 10*9/L
* Hemoglobin ≥ 9 g/dL

Hepatic:

* Total bilirubin ≤ 2 x upper limit of normal (ULN)
* Transaminases (aspartate aminotransferase (AST), serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT), serum glutamic pyruvic transaminase (SGPT) ≤ 5 x ULN

Renal:

* Creatinine clearance ≥50 mL/min based either on Cockcroft-Gault estimate or based on urine collection (12 or 24 hour)

Metabolic:

* Fasting serum glucose (≤ 130 mg/dL) and fasting triglycerides ≤ 300 mg/dL.
* Glycosylated hemoglobin (HbA1c) <7.0%

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 years or older at the time of informed consent.
* Voluntary written consent must be signed before performance of any study related procedure not part of standard medical care, with the understanding that the subject may withdraw consent at any time without prejudice to future medical care.
* Females of childbearing potential must agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 90 days after the last dose of study drug, or agree to completely abstain from heterosexual intercourse.
* Females of childbearing potential must have a negative serum pregnancy test within 7 days prior to prior to registration for protocol therapy. NOTE: Female subjects are considered of childbearing potential unless they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months.
* Male subjects, even if surgically sterilized (i.e., status post-vasectomy), must agree to practice effective barrier contraception during the entire study treatment period and through 120 days after the last dose of study drug, or agree to completely abstain from heterosexual intercourse.
* Subjects must have a diagnosis of measurable advanced or metastatic hepatocellular carcinoma (HCC). Advanced HCC is defined as disease not amenable to surgery, ablation, transplant, or embolic therapy.
* Phase II subjects must be willing to provide a tissue biopsy prior to registration if archived HCC tumor tissue is not available for correlative studies.
* For the phase I cohort, subjects with one prior systemic treatment are eligible.
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.
* Adequate organ function, as specified below, within 28 days before study registration:
* Bone marrow reserve consistent with: absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L; platelet count ≥ 50 x 10^9/L; hemoglobin ≥ 9 g/dL;
* Hepatic: total bilirubin ≤ 2 x upper limit of normal (ULN), transaminases (aspartate aminotransferase/serum glutamic oxaloacetic transaminase-AST/SGOT and alanine aminotransferase/serum glutamic pyruvic transaminase-ALT/SGPT) ≤ 5 x ULN
* Renal: creatinine clearance ≥50 mL/min based either on Cockcroft-Gault estimate or based on urine collection (12 or 24 hour);
* Metabolic: Glycosylated hemoglobin (HbA1c) ≤7.0%, fasting serum glucose (≤ 130 mg/dL) and fasting triglycerides ≤ 300 mg/dL.
* Ability to swallow oral medications.
* Measurable disease according to RECIST v1.1 and obtained by imaging within 28 days prior to registration for protocol therapy.
* Subjects who have a history of brain metastasis are eligible for the study provided all the following criteria are met:

  * Must have completed their treatment for brain metastasis
  * Must be asymptomatic
  * Must not have evidence of disease progression for ≥3 months or hemorrhage after treatment;
  * Must be off-treatment from dexamethasone for 4 weeks prior to study registration and
  * Must not have an ongoing requirement for dexamethasone or anti-epileptic drugs.
* Prior locoregional liver directed therapy is allowed as long as treatment was at least 6 weeks prior to study registration, and clear progression is demonstrated by RECIST v1.1 criteria. Subject must have recovered from the acute toxic effects (≤ grade 1 CTCAE v4) of previous anti-cancer treatment prior to study enrollment; the only exception is that grade 2 neuropathy is permitted.
* Prior radiation therapy is allowed to < 25% of the bone marrow, but is not permitted within 28 days prior to study registration.
* Estimated life expectancy > 3 months as determined by the treating physician.

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria are not to be enrolled in the study:

* Female subjects who are both lactating and breastfeeding
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Treatment with any investigational products within 28 days prior to study registration.
* No prior systemic treatment is allowed, except for subjects in the phase I cohort who are permitted one prior systemic treatment.
* Failed to recover from the reversible effects of prior anticancer therapies with the exception of alopecia and grade 2 neuropathy.
* Have initiated treatment with bisphosphonates less than 30 days prior to study registration. Concurrent bisphosphonate use is only allowed if the bisphosphonate was initiated at least 30 days prior to study registration.
* Manifestations of malabsorption due to prior gastrointestinal (GI) surgery, GI disease, or for an unknown reason that may alter the absorption of MLN0128.
* No condition that could affect the absorption of study drug, including any of the following:

  * Malabsorption syndrome
  * Disease significantly affecting gastrointestinal function
  * Bowel obstruction or sub-obstruction
* History of any of the following within the last 6 months prior to study registration:

  * Ischemic myocardial event, including angina requiring therapy and artery revascularization procedures
  * Ischemic cerebrovascular event, including transient ischemic attack (TIA) and artery revascularization procedures
  * Requirement for inotropic support (excluding digoxin) or serious (uncontrolled) cardiac arrhythmia (including atrial flutter/fibrillation, ventricular fibrillation or ventricular tachycardia)
  * Placement of a pacemaker for control of rhythm
  * New York Heart Association (NYHA) Class III or IV heart failure
  * Pulmonary embolism
* Significant active cardiovascular or pulmonary disease at the time of study registration, including:

  * Uncontrolled high blood pressure (i.e., systolic blood pressure >160 mm Hg, diastolic blood pressure > 95 mm Hg)
  * Pulmonary hypertension
  * Uncontrolled asthma or O2 saturation < 90% by ABG (Arterial Blood Gas) analysis or pulse oximetry on room air
  * Significant valvular disease; severe regurgitation or stenosis by imaging independent of symptom control with medical intervention, or history of valve replacement
  * Medically significant (symptomatic) bradycardia
  * History of arrhythmia requiring an implantable cardiac defibrillator
  * Baseline prolongation of the rate-corrected QT interval (QTc) (e.g., repeated demonstration of QTc interval > 480 milliseconds, or history of congenital long QT syndrome, or torsades de pointes)
* Initiation of treatment with hematopoietic growth factors, transfusions of blood and blood products, or systemic corticosteroids (either IV or oral steroids, excluding inhalers) within 1 week prior to study registration (subjects already receiving erythropoietin on a chronic basis for ≥ 28 days are eligible).
* Other clinically significant co-morbidities, such as uncontrolled pulmonary disease, active central nervous system disease, active infection, or any other condition that could compromise participation of the subject in the study.
* Cirrhosis with Child-Pugh score > 7
* Variceal bleeding within 1 month prior to study registration.
* Refractory encephalopathy or ascites
* Known HIV positivity
* Hepatitis B surface antigen (HBsAg) positivity without active treatment. A subject found to be HBsAg positive should be on antiviral therapy for at least two weeks prior to study registration.
* Treatment with strong inhibitors and/or inducers of cytochrome P450 (CYP) 3A4, CYP2C19 or CYP2C19 within 7 days prior to study registration.
* Subjects requiring daily or chronic use of a proton pump inhibitor (PPI) and/or having taken a PPI within 7 days prior to study registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-07-18 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2020-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathy D Miller, M.D., Principal Investigator — Big Ten Cancer Research Consortium
Locations (6):
- United States (6):
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Noth Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Penn State Cancer Institute, Hershey, Pennsylvania
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- See also: Big Ten Cancer Research Consortium Website — http://www.bigtencrc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I, Level 1: 15 mg of MLN0128: Subjects at Phase I, level 1 will receive 15mg of MLN0128 orally once weekly per dose level
- Phase I, Level 2: 20mg of MLN0128: Subjects at Phase I, level 2 will receive 20mg of MLN0128 orally once weekly per dose level
- Phase I, Level 3: 30mg of MLN0128: Subjects at Phase I, level 3 will receive 30mg of MLN0128 orally once weekly per dose level
Period: Study Treatment
Arm/Group | Phase I, Level 1: 15 mg of MLN0128 | Phase I, Level 2: 20mg of MLN0128 | Phase I, Level 3: 30mg of MLN0128
Started | 7 | 4 (This study was terminated at Phase I.) | 0 (This study was terminated at Phase I.)
Completed | 0 | 0 | 0
Not Completed | 7 | 4 | 0
Not completed — Patient Withdrawal After Therapy Start | 1 | 0 | 0
Not completed — Disease Progression | 5 | 2 | 0
Not completed — Adverse Event | 1 | 2 | 0
Period: Follow up
Arm/Group | Phase I, Level 1: 15 mg of MLN0128 | Phase I, Level 2: 20mg of MLN0128 | Phase I, Level 3: 30mg of MLN0128
Started | 7 | 4 | 0
Completed | 0 | 0 | 0
Not Completed | 7 | 4 | 0
Not completed — Death | 6 | 2 | 0
Not completed — Study Terminated | 0 | 2 | 0
Not completed — Death due to progressive disease after coming off treatment early | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This study was terminated at Phase I.The official reason for study termination was Funder Decision due to lack of accrual. Dose level 1 has 7 subjects since one of the subjects (subject #6) had to come off treatment early but did not have a DLT and so the subject was replaced to have the appropriate number of subjects for the dose decision.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I, Level 1: 15 mg of MLN0128 | Phase I, Level 2: 20mg of MLN0128 | Phase I, Level 3: 30mg of MLN0128 | Total
Number analyzed (Participants) | 7 | 4 | 0 | 11
Age, Continuous [Mean (Standard Deviation); unit: year] | 65.1 (12.6) | 64.3 (3.0) |  | 64.8 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 |  | 3
  Male | 5 | 3 |  | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 7 | 3 |  | 10
  Race: Unknown | 0 | 1 |  | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic | 1 | 0 |  | 1
  Ethnicity: Non-Hispanic | 6 | 3 |  | 9
  Ethnicity: Unknown | 0 | 1 |  | 1
ECOG PS, n(%) [Count of Participants; unit: Participants] — ECOG Performance score (0-1-2) has been collected for each subject which can be described as follows :
  0 : Fully active ; no performance restrictions.
  1 : Strenuous physical activity restricted; fully ambulatory and able to carry out light work.
  2: Capable of all self-care but unable to carry out any work activities. Up and about >50% of waking hours
  Participants
    0 | 4 | 0 |  | 4
    1 | 3 | 4 |  | 7

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD) of MLN0128
Description: The primary objective for phase I of this study is to determine the maximum tolerated dose (MTD) of MLN0128.
  Maximum Tolerated Dose is defined as the dose level at which fewer than 33% of subjects experience a dose limiting toxicity (DLT).
Time Frame: From start of treatment Day 1 (D1) until completion of two cycles of treatment (maximum 56 days)
Population: Data for this primary objective was neither collected nor analyzed due to the early termination of the study by the funder.
Arm/Group | Phase I, Level 1: 15 mg of MLN0128 | Phase I, Level 2: 20mg of MLN0128 | Phase I, Level 3: 30mg of MLN0128
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Phase II: Time to Progression (TTP)
Description: The primary endpoint of Phase II of the study is to evaluate the time to progression, which is defined as the time from randomization until tumor progression as defined by RECIST v1.1.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever occurs first, assessed up to 7 months (estimated).
Population: as for outcome 1
Groups:
- Phase II Arm A: MLN0128: Subjects randomized to experimental arm will receive MLN0128 orally at the recommended phase II dose (RP2D) once weekly.
  MLN0128 (RP2D): Phase II Arm A:
  MLN0128 administered orally at the recommended phase II dose (RP2D) once weekly.
- Phase II Arm B: Sorafenib: Subjects randomized to control arm will receive sorafenib 400mg by mouth (PO) twice a day (BID) daily.
  Sorafenib: Phase II Arm B:
  Sorafenib administered at 400mg PO BID daily
Arm/Group | Phase II Arm A: MLN0128 | Phase II Arm B: Sorafenib
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Phase I: Characterize Adverse Effects (AE)
Description: Toxicity assessed using Common Terminology Criteria for Adverse Events v4.0 (CTCAE) criteria
Time Frame: From date of first dose until 30 days after the last treatment, assessed for estimated 7 cycles (est. 196 days)
Population: This study was terminated at Phase I.The official reason for study termination was Funder Decision due to lack of accrual.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I, Level 1: 15 mg of MLN0128 | Phase I, Level 2: 20mg of MLN0128 | Phase I, Level 3: 30mg of MLN0128
Number analyzed (Participants) | 7 | 4 | 0
Participants
  Patient had at least 1 Grade 3 or greater AE | 5 | 3 |
  Patient had at least 1 Grade 3 or greater treatment related AE | 2 | 2 |
  Patient having serious adverse event | 1 | 0 |

4. Secondary Outcome: Phase I: Overall Survival (OS) Rate
Description: Overall Survival of subjects receiving MLN0128 is defined by the time from randomization to date of death from any cause.Here median overall survival in months has been reported for subjects per dose level with 95% confidence interval.
Time Frame: From date of registration until death from any cause, up to a maximum of 27 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I, Level 1: 15 mg of MLN0128 | Phase I, Level 2: 20mg of MLN0128 | Phase I, Level 3: 30mg of MLN0128
Number analyzed (Participants) | 7 | 4 | 0
months | 5.78 [2.74 to 15.68] | 10.58 [6.48 to 12.78] |

5. Secondary Outcome: Phase II: Overall Survival (OS) Rate
Description: Overall Survival of subjects randomized to both MLN0128 and sorafenib arms is defined by the time from randomization to date of death from any cause.
Time Frame: From date of registration until death from any cause, up to a maximum of 24 months
Population: as for outcome 3
Arm/Group | Phase II Arm A: MLN0128 | Phase II Arm B: Sorafenib
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Phase I: Time to Progression (TTP)
Description: Time to progression (TTP) of subjects receiving MLN0128 assessed using RECIST v1.1 criteria is defined as the time from randomization until tumor progression as defined by RECIST v1.1. Here median Time to Progression in months has been reported for subjects per dose level with 95% confidence interval.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever occurs first, assessed up to 6 months (estimated).
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I, Level 1: 15 mg of MLN0128 | Phase I, Level 2: 20mg of MLN0128 | Phase I, Level 3: 30mg of MLN0128
Number analyzed (Participants) | 7 | 4 | 0
months | 1.77 [0.57 to 1.83] | 2.83 [1.42 to 5.52] |

7. Secondary Outcome: Phase I: Progression-free Survival (PFS)
Description: Progression free survival (PFS) of subjects receiving MLN0128 assessed using RECIST v1.1 criteria is defined by time from randomization to tumor progression or death from any cause. Here median Progression-free survival in months has been reported for subjects per dose level with 95% confidence interval.
Time Frame: From date of randomization to tumor progression or death from any cause, up to a maximum of 6 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I, Level 1: 15 mg of MLN0128 | Phase I, Level 2: 20mg of MLN0128 | Phase I, Level 3: 30mg of MLN0128
Number analyzed (Participants) | 7 | 4 | 0
months | 1.81 [1.27 to 3.99] | 2.83 [1.42 to 5.52] |

8. Secondary Outcome: Phase II: Progression Free Survival (PFS)
Description: Progression Free Survival of subjects randomized to both MLN0128 and sorafenib arms assessed using RECIST v1.1 criteria, is defined as time from randomization to tumor progression or death from any cause.
Time Frame: From date of randomization to tumor progression or death from any cause, up to a maximum of 24 months
Population: as for outcome 3
Arm/Group | Phase II Arm A: MLN0128 | Phase II Arm B: Sorafenib
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Phase I: Objective Response Rate (ORR)
Description: Objective Response Rate (ORR) of subjects receiving MLN0128 defined as complete response (CR)+partial response (PR), as defined by RECIST v1.1.
Time Frame: Objective Response Rate is assessed at 16 weeks and 24 weeks from start of treatment cycle until Progressive disease is documented.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I, Level 1: 15 mg of MLN0128 | Phase I, Level 2: 20mg of MLN0128 | Phase I, Level 3: 30mg of MLN0128
Number analyzed (Participants) | 7 | 4 | 0
Participants | 0 | 0 |

10. Secondary Outcome: Phase I: Disease Control Rate (DCR)
Description: Disease Control Rate (DCR) of subjects receiving MLN0128 as a sum of stable disease (SD for 8 weeks or longer), partial response (PR), and complete response (CR), as defined by RECIST v1.1.
Time Frame: Disease Control Rate is assessed at 16 weeks and 24 weeks from start of treatment cycle until Progressive disease is documented.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I, Level 1: 15 mg of MLN0128 | Phase I, Level 2: 20mg of MLN0128 | Phase I, Level 3: 30mg of MLN0128
Number analyzed (Participants) | 7 | 4 | 0
Participants | 0 | 2 |

11. Secondary Outcome: Phase II: Characterize Adverse Effects (AE)
Description: Toxicity for subjects randomized to both MLN0128 and sorafenib arms, assessed using CTCAE v4 criteria
Time Frame: From date of first dose until 30 days after the last treatment, assessed for estimated 7 cycles (est. 196 days)
Population: as for outcome 3
Arm/Group | Phase II Arm A: MLN0128 | Phase II Arm B: Sorafenib
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Phase II: Radiographic Response Rate (RRR)
Description: Radiographic Response Rate for subjects randomized to both MLN0128 and sorafenib arms, determined utilizing objective response rate (ORR) and disease control rate (DCR) at 16 and 24 weeks.
Time Frame: Radiographic Response Rate is assessed at 16 weeks and 24 weeks from start of treatment cycle until Progressive disease is documented.
Population: as for outcome 3
Arm/Group | Phase II Arm A: MLN0128 | Phase II Arm B: Sorafenib
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded from the time of consent and for at least 30 days after treatment discontinuation, regardless of whether or not the event(s) were considered related to trial medications. Serious adverse events were reported from the initiation of study drug(s) and for 30 days after administration of the last dose of study drug(s).
Description: Adverse events were collected from the date of first treatment dose until 30 days after the last treatment, assessed for 7 cycles of treatment. Each treatment cycle was of 28 days.
Arm/Group | Phase I, Level 1: 15 mg of MLN0128 | Phase I, Level 2: 20mg of MLN0128 | Phase I, Level 3: 30mg of MLN0128
All-Cause Mortality (participants affected / at risk) | 7/7 | 2/4 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/4 | 0/0
Other Adverse Events (participants affected / at risk) | 7/7 | 4/4 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I, Level 1: 15 mg of MLN0128 (N=7) | Phase I, Level 2: 20mg of MLN0128 (N=4) | Phase I, Level 3: 30mg of MLN0128 (N=0)
GASTRIC HEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I, Level 1: 15 mg of MLN0128 (N=7) | Phase I, Level 2: 20mg of MLN0128 (N=4) | Phase I, Level 3: 30mg of MLN0128 (N=0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (3) | 2 (3) | NA
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 1 (1) | 0 (0) | NA
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1) | 0 (0) | NA
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (3) | 1 (2) | NA
ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 2 (2) | NA
ANAL FISTULA (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
ANEMIA (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | NA
ANOREXIA (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | NA
ANXIETY (Psychiatric disorders) | 2 (2) | 1 (1) | NA
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | NA
ASCITES (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 3 (4) | 3 (3) | NA
ATRIAL FIBRILLATION (Cardiac disorders) | 2 (2) | 1 (1) | NA
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | NA
BLOATING (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
BLOOD AND LYMPHATIC SYSTEM DISORDERS - OTHER, SPECIFY (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | NA
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (1) | 1 (1) | NA
BRUISING (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
CHILLS (General disorders) | 0 (0) | 1 (1) | NA
CHOLESTEROL HIGH (Investigations) | 1 (1) | 1 (1) | NA
CONFUSION (Psychiatric disorders) | 0 (0) | 1 (1) | NA
CONSTIPATION (Gastrointestinal disorders) | 4 (4) | 3 (3) | NA
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | NA
CREATININE INCREASED (Investigations) | 1 (1) | 0 (0) | NA
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0) | NA
DIARRHEA (Gastrointestinal disorders) | 4 (6) | 3 (5) | NA
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 1 (2) | NA
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | NA
DIZZINESS (Nervous system disorders) | 2 (2) | 0 (0) | NA
DYSGEUSIA (Nervous system disorders) | 1 (1) | 2 (3) | NA
DYSPHAGIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
EAR AND LABYRINTH DISORDERS - OTHER, SPECIFY (Ear and labyrinth disorders) | 0 (0) | 1 (1) | NA
EDEMA LIMBS (General disorders) | 1 (1) | 1 (2) | NA
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 0 (0) | 1 (1) | NA
EYE DISORDERS - OTHER, SPECIFY (Eye disorders) | 1 (1) | 0 (0) | NA
FATIGUE (General disorders) | 7 (9) | 4 (9) | NA
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
FEVER (General disorders) | 1 (1) | 0 (0) | NA
FLU LIKE SYMPTOMS (General disorders) | 0 (0) | 1 (1) | NA
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 (2) | 2 (2) | NA
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY (General disorders) | 1 (2) | 0 (0) | NA
GYNECOMASTIA (Reproductive system and breast disorders) | 0 (0) | 1 (1) | NA
HEADACHE (Nervous system disorders) | 2 (3) | 0 (0) | NA
HEARING IMPAIRED (Ear and labyrinth disorders) | 1 (1) | 0 (0) | NA
HEPATITIS VIRAL (Infections and infestations) | 4 (4) | 2 (2) | NA
HYPERCALCEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | NA
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 3 (4) | 4 (8) | NA
HYPERTENSION (Vascular disorders) | 5 (7) | 3 (7) | NA
HYPERTHYROIDISM (Endocrine disorders) | 1 (1) | 0 (0) | NA
HYPERURICEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | NA
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | NA
HYPONATREMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | NA
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1) | NA
HYPOKALEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | NA
HYPONATREMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | NA
HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0) | NA
IMMUNE SYSTEM DISORDERS - OTHER, SPECIFY (Immune system disorders) | 0 (0) | 1 (1) | NA
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 0 (0) | 1 (1) | NA
INSOMNIA (Psychiatric disorders) | 1 (1) | 0 (0) | NA
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 (1) | 2 (4) | NA
MUCOSITIS ORAL (Gastrointestinal disorders) | 2 (5) | 3 (7) | NA
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | NA
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA
NAUSEA (Gastrointestinal disorders) | 5 (5) | 4 (8) | NA
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | NA
NERVOUS SYSTEM DISORDERS - OTHER, SPECIFY (Nervous system disorders) | 0 (0) | 1 (1) | NA
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 2 (5) | NA
NON-CARDIAC CHEST PAIN (General disorders) | 2 (2) | 0 (0) | NA
OBESITY (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | NA
ORAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
PAIN (General disorders) | 0 (0) | 1 (1) | NA
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (2) | NA
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 (0) | 1 (1) | NA
PALPITATIONS (Cardiac disorders) | 1 (1) | 0 (0) | NA
PLATELET COUNT DECREASED (Investigations) | 2 (2) | 1 (4) | NA
PORTAL VEIN THROMBOSIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | NA
POSTNASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | NA
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | NA
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | NA
REPRODUCTIVE SYSTEM AND BREAST DISORDERS - OTHER, SPECIFY (Reproductive system and breast disorders) | 0 (0) | 1 (1) | NA
SINUS DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | NA
SLEEP APNEA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | NA
SPASTICITY (Nervous system disorders) | 0 (0) | 1 (1) | NA
TINNITUS (Ear and labyrinth disorders) | 1 (1) | 0 (0) | NA
TOOTH INFECTION (Infections and infestations) | 1 (1) | 0 (0) | NA
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 0 (0) | NA
VASCULAR DISORDERS - OTHER, SPECIFY (Vascular disorders) | 1 (1) | 1 (1) | NA
VOMITING (Gastrointestinal disorders) | 3 (5) | 0 (0) | NA
WEIGHT LOSS (Investigations) | 2 (2) | 1 (1) | NA
WHITE BLOOD CELL DECREASED (Investigations) | 0 (0) | 1 (2) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT02575339/Prot_SAP_000.pdf